CLINICAL TRIAL: NCT00261677
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Weekly PROCRIT (Epoetin Alfa) on Anemia and Quality of Life in Children With Cancer Undergoing Myelosuppressive Chemotherapy
Brief Title: A Study to Evaluate the Effect of Weekly PROCRIT (Epoetin Alfa) or Placebo on Anemia and Quality of Life in Children With Cancer Undergoing Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002296
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Hodgkin Disease; Leukemia; Lymphoma, Non-hodgkin
Keywords: Anemia; cancer; solid tumor; Hodgkin's Disease; Acute Lymphocytic Leukemia (ALL); Non-Hodgkin's Lymphoma (NHL); Quality of Life; hemoglobin; Epoetin alfa
MeSH Terms: conditions — Anemia; Hodgkin Disease; Leukemia; Lymphoma, Non-Hodgkin; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of once- weekly dosing of PROCRITÂ® (a glycoprotein that stimulates red blood cell production) versus placebo in the treatment of anemia in children with cancer undergoing chemotherapy, and to assess its effect on the quality of life.

DETAILED DESCRIPTION:
PROCRIT® (epoetin alfa) is an analogue of erythropoetin, a hormone secreted by kidneys known to stimulate red blood cell production. PROCRIT® is approved to be given three times per week to treat anemia in adult cancer patients receiving chemotherapy. Once per week dosing in adult cancer patients receiving chemotherapy is investigational and is not approved by the FDA. The use of PROCRIT® in children with cancer is investigational and is not approved by the FDA. (Please note: Since completion of this study, once weekly dosing on PROCRIT® in adult cancer patients was approved by FDA in June 2004 and use of PROCRIT® in children with cancer was approved by FDA in October 2005). The use of PROCRIT® to improve quality of life is investigational and not approved by the FDA. This is a randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of once-weekly dosing of PROCRIT® or placebo on anemia in children with cancer undergoing myelosuppressive chemotherapy, and to assess its effect on the quality of life. Patients are randomized into a 1:1 ratio to receive either PROCRIT® or placebo administered intravenously. Randomization is stratified by cancer type, with one stratum for children diagnosed with a malignant solid tumor or Hodgkin's Disease, and the second stratum for children diagnosed with Acute Lymphocytic Leukemia (ALL) or Non-Hodgkin's Lymphoma (NHL). The initial dose of study medication is 600 Units/kg for a maximum dose of 40,000 Units intravenously (IV) weekly, or placebo, up to 16 weeks. The study medication is adjusted to 900 Units/kg, for a maximum dose of 60,000 Units IV weekly, if the hemoglobin does not increase by at least 1 g/dL by Study Week 4/5. Patients were seen and evaluated based on the patient's scheduled chemotherapy regimen. Patients who received chemotherapy weekly, every two weeks, or every four weeks (4-week group), scheduled study visits occurred every four weeks. The study investigated effectiveness of once weekly dosing of PROCRIT® on anemia and quality of life in children with cancer undergoing myelosuppressive chemotherapy. The primary measure of effectiveness is the change in the patient-reported Pediatric Quality of Life Inventory (PedsQL Inventory) from baseline to the last assessment. Other measures of effectiveness include differences in hemoglobin levels, transfusion requirements, and quality of life outcomes. Safety is assessed by comparing the incidence and severity of adverse experiences in the PROCRIT® group versus the placebo group. Clinical laboratory tests (hematology, iron profile, and serum chemistry), physical examinations, and vital sign measurements are also assessed. 600 to 900 Units/kg intravenously (IV) of either PROCRIT® or placebo. Initial dose is 600 Units/kg (maximum dose 40,000 Units IV weekly) up to 16 weeks. If the hemoglobin does not increase by >= 1 g/dL at Week 4/5, dose is adjusted to 900 Units/kg (maximum dose 60,000 Units IV weekly).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed new diagnosis of malignant solid tumor, Hodgkin's disease, Acute Lymphocytic Leukemia (ALL) or Non-Hodgkin's Lymphoma (NHL)
* scheduled to receive first myelosuppressive chemotherapy within 7 days of baseline or have received up to the second myelosuppressive chemotherapy within 60 days prior to study enrollment, and scheduled to receive chemotherapy over a minimum period of 12 weeks after study enrollment
* anemic according to age-based and gender-based criteria (hemoglobin level of < 10.5 g/dL for boys and girls ages 5 to 12 years, < 11.0 g/dL for girls older than 12 years, < 12.0 g/dL for boys older than 12 years)
* have an indwelling central venous access device (e.g., subcutaneous port, external Hickman-Broviac-type catheter, or peripherally inserted central catheter) or existing peripheral intravenous catheter in place for chemotherapy administration
* both male or female patients who are reproductive potential and sexually active must be practicing an acceptable method of birth control throughout the entire study
* Parent/legal guardian must have read and signed the informed consent and patients must have provided assent, as appropriate according to state and IRB requirements

Exclusion Criteria:

* Diagnosis of myeloid leukemia or other myeloid malignancy (e.g., granulocytic sarcoma)
* diagnosis of Down's Syndrome, tumor of the central nervous system (CNS) or symptomatic metastatic CNS disease (for the solid tumor/Hodgkin's Disease stratum), or presence of symptomatic CNS disease at diagnosis (for the Acute Lymphocytic Leukemia/Non-Hodgkin's Lymphoma stratum)
* scheduled to receive cranial irradiation during the study period, or has received cranial irradiation within 30 days prior to study enrollment
* have an inherited form of anemia (hemoglobinopathy, thalassemia, red cell membrane defect, red cell enzyme deficiency) or a Coombs-positive hemolytic anemia
* elevated serum creatinine based upon age of study entry ( > 0.8 mg/dL for children younger than 10 years, > 1.1 mg/dL for children 10 - 15 years, > 1.4 mg/dL for children older than 15 years)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 224 (Actual)
Dates: Start 2000-08; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Change in the patient-reported Pediatric Quality of Life Inventory (PedsQL Inventory) from baseline to the last assessment.

SECONDARY OUTCOMES:
Parents' Quality of Life assessments on the Pediatric Quality of Life Inventory (PedsQL Inventory); Patient- and parent-reported assessments on the PedsQL Cancer Module; hemoglobin levels; transfusion requirements

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Result] Razzouk BI, Hord JD, Hockenberry M, Hinds PS, Feusner J, Williams D, Rackoff WR. Double-blind, placebo-controlled study of quality of life, hematologic end points, and safety of weekly epoetin alfa in children with cancer receiving myelosuppressive chemotherapy. J Clin Oncol. 2006 Aug 1;24(22):3583-9. doi: 10.1200/JCO.2005.03.4371. PMID 16877725
- See also: Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Weekly PROCRIT (Epoetin Alfa) on Anemia and Quality of Life in Children with Cancer Undergoing Myelosuppressive Chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=920&filename=CR002296_CSR.pdf